CLINICAL TRIAL: NCT02179515
Title: An Open Label Phase I Study to Evaluate the Safety and Tolerability of a Modified Vaccinia Ankara (MVA) Based Vaccine Modified to Express Brachyury and T-Cell Costimulatory Molecules (MVA Brachyury-TRICOM)
Brief Title: Safety and Tolerability of a Modified Vaccinia Ankara (MVA)-Based Vaccine Modified to Express Brachyury and T-cell Costimulatory Molecules (MVA-Brachyury-TRICOM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140142; 14-C-0142
Record Dates: First submitted 2014-06-28; First posted 2014-07-02 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Breast Cancer; Prostate Cancer; Tumors (Others); Ovarian Cancer
Keywords: Immune Response; Maximum Tolerated Dose; Vaccine Therapy; Increased Expression of Brachyury; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- modified vaccinia Ankara (MVA)-brachyury-TRICOM vaccine (Experimental): Three cohorts will receive modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as either 1, 2, or 4 injections of study drug at monthly (28 days +/4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
  Interventions: Biological: MVA-brachyury- TRICOM

INTERVENTIONS:
Biological: MVA-brachyury- TRICOM — It is an active cancer immunotherapy administered via subcutaneous injection.

SUMMARY:
Background:

- This cancer vaccine was developed to help teach the body's immune system to attack and destroy cancer cells. It teaches immune cells to target the Brachyury protein. This protein is present in some tumor cells, and it can help tumor cells spread to other parts of the body. Researchers want to see whether the new Brachyury protein vaccine can help treat people with advanced carcinomas.

Objective:

- To test the safety and effectiveness of giving the modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine to people with cancer.

Eligibility:

- Adults ages 18 and over whose type of cancer has not responded to standard therapies who do not have a history of autoimmune diseases and are capable of taking care of themselves.

Design:

* Participants will be screened with a medical history and physical exam. They will have blood and urine tests. They may have a computed tomography (CT) scan, a positron emission tomography (PET) scan, and a brain magnetic resonance imaging (MRI) scan. They may have a bone scan. They will have an electrocardiogram (ECG) to test heart rhythm.
* Participants will have visits about every 4 weeks. They will have a physical exam and blood and urine tests. They will be injected with the vaccine under the skin into the upper thigh or around the armpits.
* CT scans or MRI scans will be done at visit 1, after 3 months on study, and again 3 months later if still on the study. Another ECG will be done at their last vaccine visit.
* When participants stop the vaccine, they will return for visits until they recover from any side effects. They will have tests including physical exam, blood tests, scans, and x-rays.
* Participants will be asked to enroll in another study for long-term follow-up.

DETAILED DESCRIPTION:
Background:

* modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM is a novel recombinant vector-based therapeutic cancer vaccine designed to induce an enhanced immune response against brachyury, which is overexpressed in many solid tumor types, such as lung, breast, ovarian, chordoma, prostate, colorectal, and pancreatic adenocarcinoma.
* Modified vaccinia Ankara (MVA) is a replication-deficient, attenuated derivative of vaccinia. It is used in the smallpox vaccination and is now being developed as a recombinant viral vector to produce vaccines against infectious diseases and cancer.
* Many MVA vector-based trials conducted in patients with cancer have demonstrated its safety and the immunogenicity of its transgenes.
* Brachyury is a member of the T-box family of transcription factors. It is overexpressed in cancer cells compared with normal tissue and has been linked to cancer cell resistance and metastatic potential.
* Brachyury as a vaccine target has been demonstrated to be safe in an ongoing phase I study of recombinant yeast-brachyury and to generate brachyury-specific T-cell responses.
* Poxviral vaccines delivering a triad of three human T-cell costimulatory molecules designated TRICOM (B7.1, ICAM-1 and LFA-3) have been extensively studied in both preclinical and clinical studies and have demonstrated their ability to induce robust T-cell activation and provide evidence of clinical benefit.
* In vitro, MVA-brachyury-TRICOM is able to effectively expand brachyury-specific cluster of differentiation 8 (CD8+) and cluster of differentiation 4 (CD4+) T cells from peripheral blood mononuclear cells.
* Previous work indicates that MVA-brachyury-TRICOM will induce activation a distinct Tcell subpopulation from that seen with yeast-brachyury vaccine already in development.

Objectives:

To determine the safety and tolerability of escalating doses of MVA-brachyury-TRICOM vaccine.

Eligibility:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable locally advanced malignant solid tumor. In the case of chordoma, unresectable, locally recurrent, or metastatic tumors are acceptable for enrollment, given that this represents incurable disease. As much as possible, patients enrolled will have tumor types with known increased expression of brachyury (such as lung, breast, ovarian, prostate, colorectal, pancreatic, or chordoma).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at study entry
* Age greater than or equal to 18 years.
* Prior Therapy: Completed, or disease progression on at least one prior line of disease appropriate therapy for metastatic disease, or not a candidate for therapy of proven efficacy for their disease.

Design:

* This is an open-label, phase I trial with sequential cohorts of patients (3-6 patients per dose cohort) with dose escalation of MVA-brachyury-TRICOM vaccine.
* Three cohorts will receive MVA-brachyury-TRICOM vaccine administered subcutaneously as either 1, 2, or 4 injections of study drug (1 injection equal to 2 x 10^8 infectious units at monthly (28 days +/- 4 days) intervals for 3 months (treatment).
* Expansion cohorts of up to 10 patients may be enrolled at the two highest tolerated dose levels. These cohorts will allow certain standard, relatively non-toxic therapies to continue while patients receive vaccine.
* Up to 18 patients may be required to be enrolled in the 3 cohorts, plus an additional 10 at the maximum tolerated dose (MTD) and at the dose level just below it. Thus, up to 38 patients may be theoretically required to complete this trial. If 3 patients per month can be accrued, the study is expected to require 1 year to complete the necessary enrollment.

ELIGIBILITY:
* INCLUSION CRITERIA:

(All Subjects)

1. Patients must have a metastatic or unresectable locally advanced malignant solid tumor, histologically confirmed by the Laboratory of Pathology, National Cancer Institute (NCI). In the case of chordoma, unresectable, locally recurrent, or metastatic tumors are acceptable for enrollment, given that this represents incurable disease. Efforts will be made, as much as possible, to enroll patients with tumor types with known increased expression of brachyury (such as lung, breast, ovarian, prostate, colorectal, pancreatic, or chordoma; other tumors may be included as data on the level of brachyury in those tumors becomes available).
2. Patients may have measurable or nonmeasurable but evaluable disease. Patients with surgically resected metastatic disease at high risk of relapse are also eligible.
3. Prior therapy: Patients must have completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease, or not be candidates for therapy of proven efficacy for their disease.
4. There should be a minimum of 4 weeks from any prior chemotherapy, immunotherapy and/or radiation, with the exception of hormonal therapy for prostate and breast cancers, human epidermal growth factor receptor 2 (HER2)-directed therapy for HER2+ breast cancer (3+ immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH+), and erlotinib in epidermal growth factor receptor (EGFR)-mutated lung cancer in the expansion cohort as detailed in section. There should be a minimum of 6 weeks from any prior antibody therapies, (such as ipilimumab or anti-Programmed cell death protein 1 (PD1)/Programmed death-ligand 1 (PDL1) due to prolonged half-life.
5. Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy. Typically, this is 3-4 weeks for patients who most recently received cytotoxic therapy, except for the nitrosoureas and mitomycin C, for which 6 weeks is needed for recovery.
6. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
7. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 70%).
8. Patients must have normal organ and marrow function as defined below:

   * Serum creatinine less than or equal to 1.5 x upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 50 mL/min.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3 x the upper limits of normal.
   * Total bilirubin less than or equal to 1.5 x upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0.
   * Hematological eligibility parameters (within 16 days of starting therapy):

     * Granulocyte count greater than or equal to 1,500/mm^3
     * Platelet count greater than or equal to 100,000/mm^3
9. Patients must have baseline pulse oximetry > 90% on room air.
10. The effects of MVA-brachyury-TRICOM on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for a period of 4 months after the last vaccination therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. Patients with prostate cancer must continue to receive gonadotropin releasing hormone (GnRH) agonist therapy (unless orchiectomy has been done). If a patient has refused GnRH therapy, they may be enrolled on a dose level for which the safety has already been determined.

Patients must be able to understand and be willing to sign a written informed consent document.

INCLUSION CRITERIA:

(Expansion Phase Only)

The following inclusion criteria apply specifically to patients being considered for the expansion phase of the protocol.

1. Subjects with epidermal growth factor receptor (EGFR)-mutated lung cancer may continue erlotinib if they have been on the drug for greater than or equal to 3 months with stable disease or a response. Erlotinib may also be continued in the case of a progressing tumor after prior response (or > 6 months stable disease).
2. Patients with Estrogen receptor positive (ER+) breast cancer being treated with hormonal therapy (selective estrogen receptor modulator or aromatase inhibitor) who have rising tumor markers as evidence of disease progression or metastatic disease on scans may continue on hormonal therapy while being treated with vaccine.
3. Patients with Her2+ breast cancer receiving Her2-directed therapy (e.g. trastuzumab) may continue on that therapy when enrolling into a dose level for which safety has been established.
4. Subjects with metastatic colorectal cancer may continue "maintenance" therapy with capecitabine and/or bevacizumab.

EXCLUSION CRITERIA:

1. Concurrent treatment for cancer, with specific exceptions noted in inclusion criteria.
2. Chronic hepatitis B or C infection, because potential immune impairment caused by these disorders may diminish the effectiveness of this immunologic therapy.
3. Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
4. Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
5. Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. However, patients with vitiligo or clinically stable autoimmune endocrine disease who are on appropriate replacement therapy (if such therapy is indicated) are eligible.
6. Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited pharmacologic doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent intravenous (I.V.) contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.
7. Patients who are receiving any other investigational agents within 28 days before start of study treatment.
8. Patients with untreated central nervous system metastases or local treatment of brain metastases within the last 6 months. Patients with stable brain metastasis for 6 months post-intervention are eligible. Subjects with chordoma will be eligible regardless of site of disease if other eligibility criteria are met.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to MVA-brachyury-TRICOM or other agents used in study.
10. Serious or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
11. Pregnant women are excluded from this study due to the unknown effects of the MVAbrachyury-TRICOM vaccine on the fetus or infant. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MVA-brachyury-TRICOM, breastfeeding should be discontinued if the mother is treated with MVA-brachyury-TRICOM. These potential risks may also apply to other agents used in this study.
12. Human immunodeficiency viruses (HIV)-positive patients are ineligible because of the potential for decreased immune response to the vaccine.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06-28 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodge JW, Sabzevari H, Yafal AG, Gritz L, Lorenz MG, Schlom J. A triad of costimulatory molecules synergize to amplify T-cell activation. Cancer Res. 1999 Nov 15;59(22):5800-7. PMID 10582702
- [Background] Fernando RI, Litzinger M, Trono P, Hamilton DH, Schlom J, Palena C. The T-box transcription factor Brachyury promotes epithelial-mesenchymal transition in human tumor cells. J Clin Invest. 2010 Feb;120(2):533-44. doi: 10.1172/JCI38379. Epub 2010 Jan 11. PMID 20071775
- [Background] Heery CR, Palena C, McMahon S, Donahue RN, Lepone LM, Grenga I, Dirmeier U, Cordes L, Marte J, Dahut W, Singh H, Madan RA, Fernando RI, Hamilton DH, Schlom J, Gulley JL. Phase I Study of a Poxviral TRICOM-Based Vaccine Directed Against the Transcription Factor Brachyury. Clin Cancer Res. 2017 Nov 15;23(22):6833-6845. doi: 10.1158/1078-0432.CCR-17-1087. Epub 2017 Aug 30. PMID 28855356
- [Derived] Fenerty KE, Patronas NJ, Heery CR, Gulley JL, Folio LR. Resources Required for Semi-Automatic Volumetric Measurements in Metastatic Chordoma: Is Potentially Improved Tumor Burden Assessment Worth the Time Burden? J Digit Imaging. 2016 Jun;29(3):357-64. doi: 10.1007/s10278-015-9846-9. PMID 26596767

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 1 injection (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOMvaccine administered subcutaneously as 2 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 4 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
Period: Overall Study
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Started | 3 | 17 | 18
Completed | 1 | 1 | 4
Not Completed | 2 | 16 | 14
Not completed — switched to alternative treatment | 0 | 1 | 1
Not completed — Death | 0 | 1 | 1
Not completed — refused further treatment | 0 | 3 | 4
Not completed — Disease progression on study | 2 | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-modified vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 2 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU | Total
Number analyzed (Participants) | 3 | 17 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 13 | 27
  >=65 years | 0 | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (3.4) | 60.92 (11.61) | 60.31 (12.38) | 60.65 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 8 | 18
  Male | 2 | 8 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 17 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 14 | 14 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 17 | 18 | 38
Cancer Diagnosis [Count of Participants; unit: Participants]
  Chordoma | 2 | 6 | 5 | 13
  Ovarian Ca | 1 | 0 | 0 | 1
  Pancreatic Ca | 0 | 1 | 1 | 2
  Colon Ca | 0 | 5 | 4 | 9
  Lung Ca | 0 | 1 | 3 | 4
  Breast Ca | 0 | 3 | 2 | 5
  Prostate Ca | 0 | 1 | 2 | 3
  Cholangiocarcinoma | 0 | 0 | 1 | 1
Prior Treatments [Count of Participants; unit: Participants]
  1 Prior Treatment | 3 | 4 | 3 | 10
  2 Prior Treatments | 0 | 5 | 7 | 12
  3 Prior Treatments | 0 | 4 | 4 | 8
  4 Prior Treatments | 0 | 2 | 0 | 2
  5 Prior Treatments | 0 | 1 | 2 | 3
  No prior systemic therapy | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 9 months and 6 days for DL1, 17 months and 3 days for DL2, and 23 months and 13 days for DL3.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-TRICOM vaccine administered subcutaneously as 1 injection (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-TRICOM vaccine administered subcutaneously as 2 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-TRICOM vaccine administered subcutaneously as 4 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 17 | 18
Participants | 3 | 14 | 17

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: Dose-limiting toxicity (DLT) will be defined as any one of the following: Any grade ≥ 3 hematologic toxicity or grade ≥ 3 non-hematologic toxicity that is possibly, probably, or definitely related to study drug, except transient (≤ 48 hour) grade 3 fatigue, local reactions, flu-like symptoms, fever, headache, and laboratory abnormalities that are not associated with organ pathology. Also any ≥ grade 2 allergic and ≥ grade 2 autoimmune reaction(s) (except endocrine-related immune toxicity) will be defined as a DLT. Any grade 3 autoimmune endocrine-related toxicity that has not resolved clinically within 7 days of initiating therapy will also be defined as a DLT. Generalized erythroderma or macular or papular rash lasting less than 7 days and not associated with desquamation will not be DLTs.
Time Frame: 28 days following the first injection of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 17 | 18
Participants | 0 | 0 | 0

3. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD will be the dose level at which no greater than 1/6 patients have a dose-limiting toxicity (DLT), and the next higher dose level has at least 2 patients with a DLT.
Time Frame: First 28 days of treatment.
Measure: Number; unit: 10^8 IU
Groups:
- All Participants: All participants in Dose Level 1 - 1 injection - Total Dose 2 x 10^8 IU, Dose Level 2 - 2 injections - Total Dose 4 x 10^8 IU, and Dose Level 3 - 4 injections - Total Dose 8 x 10^8 IU.
Arm/Group | All Participants
Number analyzed (Participants) | 38
10^8 IU | NA — The MTD was not reached.

4. Primary Outcome: Number of Participants With Grade 3 or Greater Adverse Events Possibly Related to Vaccine
Description: Number of participants with Grade 3 or greater adverse events possibly related to vaccine assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe or medically significant but not immediately life-threatening. Grade 4 is life threatening consequences, and Grade 5 is death related to adverse event.
Time Frame: as for outcome 1
Population: Only one Grade 3 adverse event (diarrhea) possibly related to vaccine occurred on this trial; and no Grade 4 and 5 adverse events possibly related to vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 17 | 18
Participants | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Brachyury-Specific T-cell Responses Developed After 1, 2, and 3 Vaccinations
Description: A fluorescence activated cell sorting (FACS)-based assay for cluster of differentiation 4 (CD4) or cluster of differentiation 8 (CD8) T-cells expressing the cytokines interferon (IFN) gamma, interleukin 2 (IL2), and tumor necrosis factor (TNF) alpha, and/or cluster of differentiation 107a (CD107a) (a marker for lytic potential) was used to determine the numbers of participants showing development or enhancement of the level of brachyury-specific T-cells after vaccination.
Time Frame: Baseline (pre-vaccination), approximately day 29 (after 1 vaccination), approximately day 57 (after 2 vaccinations), and approximately day 85 (after 3 vaccinations)
Population: Sufficient peripheral blood mononuclear cells (PBMCs) were available before and after vaccination from 34 of 38 patients to analyze brachyury-specific CD4 and CD8 T-cell responses.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 15 | 16
Participants
  CD107a + CD4 T-cell response (d29 vs pre) | 0 | 4 | 0
  IFN gamma + CD4 T-cell response (d29 vs pre) | 1 | 2 | 1
  IL2 + CD4 T-cell response (d29 vs pre) | 1 | 1 | 0
  TNF alpha + CD4 T-cell response (d29 vs pre) | 0 | 4 | 0
  CD107a + CD8 T-cell response (d29 vs pre) | 1 | 1 | 0
  IFN gamma + CD8 T-cell response (d29 vs pre) | 0 | 6 | 0
  IL2 + CD8 T-cell response (d29 vs pre) | 0 | 0 | 0
  TNF alpha + CD8 T-cell response (d29 vs pre) | 1 | 4 | 0
  Any T-cell response (d29 vs pre) | 1 | 9 | 6
  CD107a + CD4 T-cell response (d57 vs pre) | 0 | 3 | 0
  IFN gamma + CD4 T-cell response (d57 vs pre) | 0 | 0 | 0
  IL2 + CD4 T-cell response (d57 vs pre) | 0 | 1 | 0
  TNF alpha + CD4 T-cell response (d57 vs pre) | 0 | 0 | 0
  CD107a + CD8 T-cell response (d57 vs pre) | 0 | 3 | 0
  IFN gamma + CD8 T-cell response (d57 vs pre) | 0 | 2 | 0
  IL2 + CD8 T-cell response (d57 vs pre) | 0 | 0 | 0
  TNF alpha + CD8 T-cell response (d57 vs pre) | 0 | 5 | 0
  Any T-cell response (d57 vs pre) | 0 | 6 | 10
  CD107a + CD4 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  CD107a + CD4 T-cell response (d85 vs pre) | 0 | 2 | 0
  IFN gamma + CD4 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  IFN gamma + CD4 T-cell response (d85 vs pre) | 0 | 1 | 0
  IL2 + CD4 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  IL2 + CD4 T-cell response (d85 vs pre) | 0 | 3 | 0
  TNF alpha + CD4 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  TNF alpha + CD4 T-cell response (d85 vs pre) | 0 | 1 | 0
  CD107a + CD8 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  CD107a + CD8 T-cell response (d85 vs pre) | 0 | 2 | 0
  IFN gamma + CD8 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  IFN gamma + CD8 T-cell response (d85 vs pre) | 0 | 0 | 0
  IL2 + CD8 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  IL2 + CD8 T-cell response (d85 vs pre) | 0 | 0 | 0
  TNF alpha + CD8 T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  TNF alpha + CD8 T-cell response (d85 vs pre) | 0 | 1 | 0
  Any T-cell response (d85 vs pre): number analyzed (Participants) | 3 | 14 | 15
  Any T-cell response (d85 vs pre) | 0 | 5 | 9

6. Secondary Outcome: Percentage of Total Peripheral Blood Mononuclear Cells (PBMCs) in Peripheral Blood Before Vaccination, and After 1 and 3 Vaccinations
Description: Blood samples collected were analyzed by multicolor flow cytometry in PBMCs for cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), Natural Killer (NK), Natural Killer T (NKT), conventional dendritic cell (cDC), plasmacytoid dendritic cell (pDC), myeloid-derived suppressor cell (MDSC) and Tregs. Changes in levels PBMC subsets was a descriptive result with median and interquartile range reported. No formal statistical analysis by dose level was performed given the small sample size.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination) and D85 (post 3 vaccinations)
Population: Sufficient peripheral blood mononuclear cells (PBMCs) were available before and after vaccination from 36 of 38 patients to analyze peripheral immune cell subsets.
Measure: Median (Inter-Quartile Range); unit: Percentage of Total PBMC's
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 16 | 17
Percentage of Total PBMC's
  CD4 Pre | 24.31 [14.78 to 38.24] | 32.64 [27.63 to 40.74] | 32.89 [22.61 to 37.37]
  CD4 D29 | 23.68 [13.15 to 36.09] | 34.99 [23.61 to 39.35] | 29.86 [20.99 to 36.08]
  CD4 D85: number analyzed (Participants) | 3 | 14 | 15
  CD4 D85 | 27.70 [13.09 to 39.84] | 30.35 [25.55 to 36.67] | 29.87 [25.77 to 36.65]
  CD8 Pre | 7.51 [4.90 to 14.31] | 16.85 [10.20 to 23.58] | 12.27 [9.28 to 16.34]
  CD8 D29 | 7.83 [3.73 to 13.43] | 16.28 [9.55 to 24.45] | 10.96 [9.18 to 17.43]
  CD8 D85: number analyzed (Participants) | 3 | 14 | 15
  CD8 D85 | 10.92 [5.71 to 13.99] | 17.17 [12.29 to 26.14] | 13.99 [11.78 to 20.43]
  Treg Pre | 2.19 [1.00 to 2.41] | 1.50 [1.21 to 1.93] | 1.07 [0.77 to 1.53]
  Treg D29 | 1.71 [1.23 to 1.98] | 1.40 [1.20 to 1.78] | 1.34 [0.88 to 1.65]
  Treg D85: number analyzed (Participants) | 3 | 14 | 15
  Treg D85 | 2.09 [1.19 to 2.30] | 1.26 [0.80 to 1.65] | 1.22 [0.74 to 1.63]
  B cells Pre | 15.89 [10.45 to 21.33] | 7.76 [5.32 to 15.31] | 10.41 [6.20 to 12.44]
  B cells D29 | 15.46 [10.50 to 20.42] | 7.52 [5.54 to 15.24] | 8.56 [6.55 to 11.97]
  B cells D85: number analyzed (Participants) | 3 | 14 | 15
  B cells D85 | 14.54 [12.17 to 16.91] | 6.49 [5.32 to 11.82] | 10.26 [6.30 to 14.01]
  NK cells Pre | 6.47 [5.35 to 8.33] | 6.07 [4.23 to 9.07] | 8.93 [4.74 to 13.82]
  NK cells D29 | 7.51 [5.40 to 8.28] | 7.32 [5.82 to 11.97] | 12.34 [6.90 to 18.94]
  NK cells D85: number analyzed (Participants) | 3 | 14 | 15
  NK cells D85 | 10.30 [6.98 to 18.52] | 7.83 [6.50 to 9.57] | 12.29 [7.55 to 14.45]
  NK-T cells Pre | 0.29 [0.24 to 0.52] | 1.69 [1.20 to 5.93] | 1.90 [1.00 to 2.78]
  NK-T cells D29 | 0.35 [0.31 to 0.55] | 2.06 [0.95 to 6.09] | 2.23 [0.85 to 2.75]
  NK-T cells D85: number analyzed (Participants) | 3 | 14 | 15
  NK-T cells D85 | 0.42 [0.25 to 0.43] | 2.14 [0.94 to 6.48] | 2.03 [0.74 to 2.91]
  cDC Pre | 0.24 [0.22 to 0.58] | 0.23 [0.13 to 0.31] | 0.27 [0.20 to 0.40]
  cDC D29 | 0.46 [0.27 to 0.54] | 0.18 [0.12 to 0.27] | 0.22 [0.17 to 0.35]
  cDC D85: number analyzed (Participants) | 3 | 14 | 15
  cDC D85 | 0.28 [0.14 to 0.52] | 0.18 [0.15 to 0.24] | 0.22 [0.16 to 0.32]
  pDC Pre | 0.13 [0.12 to 0.25] | 0.15 [0.10 to 0.22] | 0.17 [0.10 to 0.36]
  pDC D29 | 0.16 [0.15 to 0.24] | 0.17 [0.11 to 0.21] | 0.22 [0.12 to 0.36]
  pDC D85: number analyzed (Participants) | 3 | 14 | 15
  pDC D85 | 0.07 [0.07 to 0.39] | 0.15 [0.12 to 0.21] | 0.23 [0.14 to 0.30]
  MDSC Pre | 13.17 [6.84 to 19.50] | 7.11 [4.86 to 10.69] | 7.04 [4.92 to 10.18]
  MDSC D29 | 8.53 [6.42 to 10.63] | 6.69 [4.27 to 11.29] | 7.66 [4.91 to 10.54]
  MDSC D85: number analyzed (Participants) | 3 | 14 | 15
  MDSC D85 | 8.34 [6.52 to 10.16] | 9.15 [5.11 to 11.94] | 8.83 [4.58 to 11.42]

7. Secondary Outcome: Number of Participants With Positive Anti-Brachyury Antibodies
Description: A positive brachyury antibody titer consisted of an absorbance to brachyury protein that was twice that obtained with the negative control protein Bovine serum albumin (BSA). A positive titer after vaccination may be indicative of an immune response to the vaccine.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination), D57 (post 2 vaccinations) and D85 (post 3 vaccinations)
Population: Sufficient serum was available before and after vaccination from 34 of 38 patients to analyze anti-brachyury antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 15 | 16
Participants
  Anti-Brachyury Antibodies Pre | 0 | 1 | 2
  Anti-Brachyury Antibodies D29 | 0 | 1 | 3
  Anti-Brachyury Antibodies D57: number analyzed (Participants) | 3 | 14 | 16
  Anti-Brachyury Antibodies D57 | 0 | 1 | 5
  Anti-Brachyury Antibodies D85: number analyzed (Participants) | 3 | 14 | 15
  Anti-Brachyury Antibodies D85 | 0 | 1 | 4

8. Secondary Outcome: Changes in Serum Cytokines Soluble CD27 (sCD27) and Soluble Factors
Description: Serum levels of Soluble CD27 (sCD27) were determined by enzyme-linked immunosorbent assay (ELISA) pre and post vaccination. Changes in levels of serum cytokines and soluble factors was a descriptive result with median and interquartile range reported. No formal statistical analysis by dose level was performed given the small sample size.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination), and D85 (post 3 vaccinations)
Population: Sufficient serum was available before and after vaccination from 36 of 38 patients to analyze serum cytokines and soluble factors.
Measure: Median (Inter-Quartile Range); unit: U/mL
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 16 | 17
U/mL
  sCD27 Pre | 20.53 [1.20 to 51.33] | 19.34 [11.24 to 23.57] | 12.10 [7.42 to 18.88]
  sCD27 D29 | 25.65 [16.30 to 47.38] | 18.40 [8.02 to 27.10] | 15.12 [11.95 to 25.82]
  sCD27 D85: number analyzed (Participants) | 3 | 14 | 15
  sCD27 D85 | 22.35 [19.03 to 24.15] | 14.50 [9.06 to 25.38] | 16.33 [12.10 to 25.99]

9. Secondary Outcome: Changes in Serum Cytokines Soluble CD40 Ligand (sCD40L) and Soluble Factors
Description: Serum levels of sCD40L, were determined by enzyme-linked immunosorbent assay (ELISA) pre and post vaccination. Changes in levels of serum cytokines and soluble factors was a descriptive result with median and interquartile range reported. No formal statistical analysis by dose level was performed given the small sample size.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination), and D85 (post 3 vaccinations)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 16 | 17
ng/mL
  sCD40L Pre | 4.76 [1.55 to 20.34] | 17.52 [11.98 to 22.03] | 18.94 [14.63 to 26.29]
  sCD40L D29 | 17.11 [1.00 to 19.79] | 17.81 [14.92 to 20.27] | 16.05 [11.25 to 19.85]
  sCD40L D85: number analyzed (Participants) | 3 | 14 | 15
  sCD40L D85 | 10.33 [1.40 to 18.35] | 17.54 [9.77 to 20.32] | 17.90 [14.03 to 21.75]

10. Secondary Outcome: Changes in the Ratio of Serums Soluble CD27 (sCD27):Soluble CD40 Ligand (sCD40L)
Description: Serum levels of sCD27, sCD40L, and the ratio of sCD27:sCD40L were determined by enzyme-linked immunosorbent assay (ELISA) pre and post vaccination. Changes in levels of serum cytokines and soluble factors was a descriptive result with median and interquartile range reported. No formal statistical analysis by dose level was performed given the small sample size.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination), and D85 (post 3 vaccinations)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 16 | 17
Ratio
  sCD27:sCD40L Pre | 4.31 [0.06 to 33.06] | 1.02 [0.56 to 1.94] | 0.64 [0.35 to 1.28]
  sCD27:sCD40L D29 | 1.50 [0.82 to 47.38] | 1.25 [0.42 to 2.06] | 0.82 [0.59 to 2.13]
  sCD27:sCD40L D85: number analyzed (Participants) | 3 | 14 | 15
  sCD27:sCD40L D85 | 1.84 [1.22 to 17.28] | 1.05 [0.53 to 2.71] | 0.89 [0.69 to 1.47]

11. Secondary Outcome: Changes in Serum Cytokines Interleukin 2 (IL2), Interleukin 4 (IL4), Interleukin 10 (IL10), and Interferon Gamma (IFNg)
Description: Serum levels of IL-2, IL-4, IL-10, and IFNg were determined by enzyme-linked immunosorbent assay (ELISA) pre and post vaccination. Changes in levels of serum cytokines and soluble factors was a descriptive result with median and interquartile range reported. No formal statistical analysis by dose level was performed given the small sample size.
Time Frame: Pre (Baseline), and approximately D29 (Post 1 vaccination), and D85 (post 3 vaccinations)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 3 | 16 | 17
pg/mL
  IL-2 Pre | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-2 D29 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-2 D85: number analyzed (Participants) | 3 | 14 | 15
  IL-2 D85 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-10 Pre | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-10 D29 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-10 D85: number analyzed (Participants) | 3 | 14 | 15
  IL-10 D85 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-4 Pre | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-4 D29 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IL-4 D85: number analyzed (Participants) | 3 | 14 | 15
  IL-4 D85 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  IFNg Pre: number analyzed (Participants) | 3 | 14 | 15
  IFNg Pre | 1.42 [0.00 to 26.11] | 0.16 [0.06 to 1.42] | 1.23 [0.00 to 94.87]
  IFNg D29 | 1.23 [0.00 to 31.59] | 0.84 [0.26 to 2.17] | 0.74 [0.00 to 131.90]
  IFNg D85: number analyzed (Participants) | 3 | 14 | 15
  IFNg D85 | 1.13 [0.16 to 28.90] | 0.55 [0.26 to 2.10] | 1.62 [0.00 to 130.20]

12. Other Pre Specified Outcome: Correlation of Brachyury Expression in Tissue Samples With Clinical Outcomes.
Description: Correlation of brachyury expression in tissue samples with clinical outcomes.
Time Frame: 2 -3 years
Population: Tissue collection was optional and insufficient tissue was obtained to perform this analysis.
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 9 months and 6 days for DL1, 17 months and 3 days for DL2, and 23 months and 13 days for DL3.
Groups:
- Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 1 injection (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 2 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
- Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU: Participants received Modified Vaccinia Ankara (MVA)-brachyury-B7-1, ICAM-1 (Intercellular Adhesion Molecule 1), and LFA-3 (lymphocyte function-associated antigen 3) TRICOM vaccine administered subcutaneously as 4 injections (I injection = 2 x 10^8 IU) of study drug at monthly (28 days +/- 4 days) intervals for 3 months. Patients with stable disease may continue to receive vaccine for up to 6 monthly doses.
Arm/Group | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/17 | 1/18
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/17 | 2/18
Other Adverse Events (participants affected / at risk) | 3/3 | 14/17 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU (N=3) | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU (N=17) | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU (N=18)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 1 Injection - Total Dose 2 x 10^8 IU (N=3) | Dose Level 2 - 2 Injections - Total Dose 4 x 10^8 IU (N=17) | Dose Level 3 - 4 Injections - Total Dose 8 x 10^8 IU (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 2 (3) | 13 (21) | 15 (34)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Fever (General disorders) | 2 (4) | 0 (0) | 6 (7)
Flu like symptoms (General disorders) | 3 (3) | 0 (0) | 12 (20)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, elevated neutrophil count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02179515/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02179515/ICF_001.pdf